CLINICAL TRIAL: NCT06904859
Title: The Role and Mechanism of TCR-T Cells in Immunotherapy for Acute Myeloid Leukemia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shenzhen University General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEM-ONCO-029
Record Dates: First submitted 2025-03-12; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Hematologic Diseases; Leukemia; Leukemia, Myeloid; TCR gene-modified T cells; immunotherapy; TCR-T cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Hematologic Diseases; Leukemia; Leukemia, Myeloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AML patients group (Experimental): To construct TCR sequence database of acute myeloid leukemia patients, and then to verify the effect and mechanism of immunotherapy in vitro and in mice，then TCR gene-modified T cells were infused back into the patients
  Interventions: Biological: TCR-T Cells Injection

INTERVENTIONS:
Biological: TCR-T Cells Injection — The TCR sequences of AML patients were analyzed by next generation sequencing to find the specific TCR clone against leukemia，then TCR gene-modified T cells were infused back into the patients

SUMMARY:
Acute myeloid leukemia (AML) is the main type of leukemia, accounting for about 60% of all leukemia, with complex pathogenesis and great clinical heterogeneity. Effective targets for AML need to be further developed. We performed next-generation sequencing analysis of the TCR sequence of an AML patient to find the patient's specific TCR clone for leukemia. The rearranged TCR gene stimulated by leukemia antigens was transduced into the patient's own T cells, and the TCR gene-modified T cells (TCR-T) that could specifically recognize leukemia antigens and kill leukemia cells were constructed. Enhancing the specificity and killing activity of T cells can truly achieve individualized treatment for patients. In addition, through TCR sequencing, the TCR sequence database of leukemia patients can be constructed to find the common specific TCR clones for AML among different patients, which can realize the precise treatment of AML.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is the main type of leukemia, accounting for about 60% of all leukemia, with complex pathogenesis and great clinical heterogeneity. Effective targets for AML need to be further developed. T cell receptor (TCR) is a characteristic marker on the surface of T cells. Stimulated by leukemia cell antigens, TCR can produce specific rearrangement and produce specific T cell clones for leukemia. However, immunosuppressive cells and immunosuppressive molecules in the leukemia microenvironment have inhibitory effects on T cells, which reduce the activity of T cells with specific clone proliferation. The anti-tumor effect was weakened. In order to solve this clinical problem, we performed next-generation sequencing analysis of the TCR sequence of an AML patient to find the patient's specific TCR clone against leukemia. The rearranged TCR gene stimulated by leukemia antigen was transduced into the patient's own T cells. To construct TCR gene-modified T cells (TCR-T) that can specifically recognize leukemia antigens and kill leukemia cells, enhance the specificity and killing activity of T cells, and truly realize the individualized treatment of patients. In addition, through TCR sequencing, the TCR sequence database of leukemia patients can be constructed to find the common specific TCR clones for AML among different patients, which can realize the precise treatment of AML.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 (≥ 18 years old, ≤ 65 years old)
2. gender is not limited
3. Acute myeloid leukemia patients
4. CR(remission phase, white blood cell count > 2×10^9/L after blood picture recovery)
5. After 3-4 courses of chemotherapy (the number of courses is not absolute)
6. Before the next chemotherapy

Exclusion Criteria:

1. Transformed acute myeloid leukemia
2. Secondary acute myeloid leukemia
3. Post-transplantation acute myeloid leukemia
4. AML-M3
5. white blood cell count <2×10^9/L
6. More than 8 courses of chemotherapy
7. Combined with other immune-related diseases
8. Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Decreased AML percentage in blood | From date of initial treatment to the 20 days after TCR-T Cells infusion
  TCR-T Cells were infused back into the patients then the decreased percentage of AML tumor cells in blood after infusion was measured

SECONDARY OUTCOMES:
Decreased AML percentage in cerebrospinal fluid | From date of initial treatment to the 20 days after TCR-T Cells infusion
  TCR-T Cells were infused back into the patient then the decreased percentage of AML tumor cells in cerebrospinal fluid after infusion was measured

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen University General Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No